CLINICAL TRIAL: NCT04152824
Title: Behavioral Health & Resilience Training for Military Leaders
Brief Title: Readiness Supportive Leadership Training
Acronym: RESULT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland State University (Other)
Responsible Party: Principal Investigator, Leslie Hammer, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: W81XWH-18-PHTBIRP-R2OE-TRA
Record Dates: First submitted 2019-10-18; First posted 2019-11-05 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Health Behavior; Well-Being
Keywords: Psychological Health; Well-Being; Resilience; Readiness; Military; Service Member
MeSH Terms: conditions — Health Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group Units (Experimental): Units randomized to the intervention group will go through the Resilience-Supportive Leadership Training (RESULT)
  Interventions: Behavioral: Resilience-Supportive Leadership Training (RESULT)
- Control Group (No Intervention): Units randomized to the control group will be usual practice regarding resiliency training

INTERVENTIONS:
Behavioral: Resilience-Supportive Leadership Training (RESULT) — Platoon leaders receive a 90-minute, in-person training addressing supportive supervisor behaviors and resilience
  Arms: Training Group Units

SUMMARY:
This study is a randomized controlled trial that assesses the effects of an evidence based, multi-component, leadership support intervention, Resilience-Supportive Leadership Training (RESULT), using accelerated learning strategies aimed at improving Service Member resilience and readiness in the military.

The intervention is expected to increase perceptions of resilience-supportive behaviors, resilience indicators, and related behavioral health outcomes such as emotion regulation, connectedness, team cohesion, and psychological health following the training from the perspective of the Service Member.

DETAILED DESCRIPTION:
The goal of our proposed study is to adapt our existing, evidence-based supportive leadership training for an active duty population, focusing on training junior leaders in the Army on ways they can enhance readiness and resilience in their soldiers, as well as their own resilience. The investigators draw on best practices from existing military and civilian programs in a training that is engaging, interactive, and customizable. The investigators use micro-learnings - small, bite-sized pieces of information delivered in non-traditional ways, such as short podcasts or videos to enhance the training and enable it to be integrated easily into both military and civilian jobs.

The investigators evaluate the effectiveness of our Resilience-Supportive Leadership Training (RESULT) intervention with U.S. Army soldiers stationed at Joint Base Lewis-McChord (JBLM) in the State of Washington. The study includes a control group, so the investigators can better determine whether any observed changes in our participants are due to our training programs, and not some other factor. The investigators anticipate that the training programs will have a positive impact on service member readiness and resilience, psychological health, team cohesion, and reduced loneliness.

This research is designed to benefit not only U.S. Army soldiers but across all military branches, as well as first-responders and other civilian occupations that face highly stressful situations as part of their work. Our training has the potential to positively contribute to the military by enhancing service member readiness and unit autonomy, and improving mental and physical health.

ELIGIBILITY:
Inclusion Criteria:

Active Duty Service Members Serving in one of the two Striker Brigade Combat Teams (SBCT).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1890 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2025-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hammer, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Joint Base Lewis McChord, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohr C, Hammer L, Dimoff J, Allen S, Lee J, Arpin S, McCabe S, Brockwood K, Bodner T, Mahoney L, Dretsch M, Britt T. Supportive-leadership training to improve social connection: A cluster-randomized trial demonstrating efficacy in a high-risk occupational context. J Occup Health Psychol. 2024 Oct;29(5):299-316. doi: 10.1037/ocp0000384. Epub 2024 Aug 15. PMID 39146072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of Service Members at all levels within the participating Battalions occurred during the month of September 2019. An Operations Order was delivered to Battalion leaders to send out an email, created by the research team, which explained the study, that participation was voluntary and confidential, and provided a link to an online survey. These emails were forwarded from the Battalion leadership to lower ranking leaders, who then sent to their individual unit members.
Pre-assignment Details: No participants who were enrolled were excluded from the study before assignment to groups.
Units Other Than Participants: Battalion
Groups:
- Service Member in Battalion Randomized to Intervention Condition: Military service members who are in a battalion randomized to the intervention condition.
- Service Member in Battalion Randomized to Control Condition: Military service members who are in a battalion randomized to the control condition.
Period: Overall Study
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Started | 948; 5 Battalion | 942; 5 Battalion
Completed | 118; 5 Battalion | 158; 5 Battalion
Not Completed | 830; 0 Battalion | 784; 0 Battalion

BASELINE CHARACTERISTICS:
Population: Service members in a randomized battalion
Groups:
- Service Member in Battalion Randomized to Intervention Condition: Military service members who are in a battalion randomized to the intervention condition. The Platoon Leaders of service members in this condition were assigned to completed the Readiness Supportive Leadership Training (RESULT).
- Service Member in Battalion Randomized to Control Condition: Military service members who are in a battalion randomized to the control condition. The Platoon Leaders of service members in this condition were assigned to usual practice.
- Total: Total of all reporting groups
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition | Total
Number analyzed (Participants) | 118 | 158 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (4.42) | 24.4 (5.01) | 23.9 (4.70)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data/responses
  Participants
    number analyzed (Participants) | 114 | 152 | 266
    Female | 100 | 144 | 244
    Male | 14 | 8 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Only high level race/ethnicity information provided for categories that are non-White as cells were so small as to potentially compromise confidentiality.
  Participants
    White & Non-White/Multiple: White | 58 | 83 | 141
    White & Non-White/Multiple: Non-White/Multiple selected/Missing | 60 | 75 | 135
Region of Enrollment [Number; unit: participants]
  United States | 118 | 158 | 276
Loneliness [Mean (Standard Deviation); unit: units on a scale] — Brief Loneliness Scale, 3 items, response options: 1 = Never 2 = Rarely 3 = Sometimes 4 = Always, summed score, range from 4-12.
  Higher score indicates higher levels of loneliness.
  Hughes, M. E., Waite, L. J., Hawkley, L. C., & Cacioppo, J. T. (2004). A short scale for measuring loneliness in large surveys: Results from two population-based studies. Research on aging, 26(6), 655-672. https://doi.org/10.1177/0164027504268574
  units on a scale | 6.44 (2.64) | 6.45 (2.58) | 6.45 (2.60)
Dimensions of Anger (DAR-5) [Mean (Standard Deviation); unit: units on a scale] — Dimensions of Anger (DAR-5), 5 items, response options: 1 = None of the time 2 = A little of the time 3 = Some of the time 4 =Most of the time 5 = All of the time, Mean score, range 1-5, with higher scores indicating higher levels of anger.
  Forbes, D., Alkemade, N., Hopcraft, D., Hawthorne, G., O'Halloran, P., Elhai, J. D., … Lewis, V. (2014). Evaluation of the Dimensions of Anger Reactions-5 (DAR-5) Scale in combat veterans with posttraumatic stress disorder. Journal of Anxiety Disorders, 28(8), 830-835. https://doi.org/10.1016/j.janxdis.2014.09.015
  units on a scale | 1.62 (.69) | 1.79 (.86) | 1.71 (.79)
Emotional Support from Leader [Mean (Standard Deviation); unit: units on a scale] — Leader Emotional Support, 3 items, response options: 1 = Strongly disagree 2 = Disagree 3 = Neither agree nor disagree 4 = Agree 5 = Strongly agree, Mean score, range 1-5, with higher scores indicating higher levels of leadership emotional support.
  Created specifically for this study based on training content.
  units on a scale | 3.88 (.91) | 4.01 (.97) | 3.95 (.95)
Life Satisfaction [Mean (Standard Deviation); unit: units on a scale] — Satisfaction with Life Scale, 5 items, response options: 1 = Strongly disagree 2 = Disagree 3 = Neither agree nor disagree 4 = Agree 5 = Strongly agree. Mean score created with range from 1-5, with higher scores indicating higher levels of life satisfaction.
  Diener, E. D., Emmons, R. A., Larsen, R. J., & Griffin, S. (1985). The satisfaction with life scale. Journal of Personality Assessment, 49(1), 71-75.
  units on a scale | 3.26 (1.00) | 3.15 (1.11) | 3.19 (1.06)
Unit Belongingness [Mean (Standard Deviation); unit: units on a scale] — Team Cohesion, Belonging Subscale, 3 items, response options: 1 = Strongly disagree 2 = Moderately disagree 3 = Slightly disagree 4 = Neither agree nor disagree 5 = Slightly agree 6 = Moderately agree 7 = Strongly agree. Mean score calculated, range 1-7, with higher scores indicating greater belonging to the unit.
  Chin, W. W., Salisbury, W. D., Pearson, A. W., & Stollak, M. J. (1999). Perceived cohesion in small groups: Adapting and testing the perceived cohesion scale in a small-group setting. Small group research, 30(6), 751-766. https://doi.org/10.1177/104649649903000605
  units on a scale | 5.45 (1.75) | 5.63 (1.65) | 5.53 (1.69)

OUTCOME MEASURES:

1. Primary Outcome: Resilience Supportive Supervisor Behaviors - Emotional Support
Description: Service member's perceptions of leadership emotional support behavior. Likert-type scale 1-5, with higher scores indicating greater support
Time Frame: 3-month post intervention, up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Number analyzed (Participants) | 118 | 158
score on a scale | 4.00 (.92) | 3.90 (1.06)

2. Primary Outcome: Resilience Supportive Supervisor Behaviors - Destigmatizing
Description: Service member's perceptions of leadership support behavior in destigmatizing behavioral health. Likert-type scale 1-5, with higher scores indicating greater destigmatization
Time Frame: 3-month post intervention, up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Number analyzed (Participants) | 118 | 158
score on a scale | 4.03 (.86) | 3.94 (1.03)

3. Primary Outcome: Dimensions of Anger Reactions (DAR-5)
Description: Service member's perceptions of their anger, Likert-type scale 1-5 with higher scores indicating higher levels of anger
Time Frame: 3-month post intervention, up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Number analyzed (Participants) | 118 | 158
score on a scale | 1.51 (.66) | 1.71 (.84)

4. Primary Outcome: Life Satisfaction
Description: Service member's perceptions of their general life satisfaction. Likert-type scale from 1-5, with higher scores indicating higher satisfaction
Time Frame: 3-month post intervention, up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Number analyzed (Participants) | 118 | 158
score on a scale | 3.23 (1.04) | 3.13 (.98)

5. Primary Outcome: Unit Belonging - Subscale of the Team Cohesion Scale
Description: Service member's perceptions degree to which they feel part of their current platoon. Likert-type scale from 1-7, with higher scores indicating more sense of belonging.
Time Frame: 3-month post intervention, up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Number analyzed (Participants) | 118 | 158
score on a scale | 5.69 (1.6) | 5.36 (1.81)

6. Primary Outcome: Brief Loneliness Scale
Description: Service member's perception of their own loneliness. Likert-type scale from 3-13, with higher scores indicating greater loneliness
Time Frame: 3-month post intervention, up to 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
Number analyzed (Participants) | 118 | 158
score on a scale | 6.21 (2.62) | 6.53 (2.74)

ADVERSE EVENTS:
Time Frame: Data collected over 6 months
Description: Study was minimal risk
Arm/Group | Service Member in Battalion Randomized to Intervention Condition | Service Member in Battalion Randomized to Control Condition
All-Cause Mortality (participants affected / at risk) | 0/948 | 0/942
Serious Adverse Events (participants affected / at risk) | 0/948 | 0/942
Other Adverse Events (participants affected / at risk) | 0/948 | 0/942

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT04152824/Prot_SAP_000.pdf